CLINICAL TRIAL: NCT05932472
Title: Randomized Comparison of Morning Versus Bedtime Administration of Aspirin: A Cardiovascular Circadian Chronotherapy (C3) Trial
Acronym: ASPIRIN-C3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, MD, MSc, MPH, PhD, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASPIRIN-C3
Record Dates: First submitted 2023-06-22; First posted 2023-07-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Drug Effect
Keywords: Aspirin; Cardiovascular Disease; Prevention; Circadian Rhythm; Randomized Controlled Trial; Pragmatic; Outcomes
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin at bedtime (Experimental): Participants randomized to aspirin administration at bedtime will be instructed to take their aspirin at approx. 8PM-12AM.
  Interventions: Drug: Aspirin
- Aspirin in the morning (Active Comparator): Participants randomized to aspirin administration in the morning will be instructed to take their aspirin upon awakening or with their breakfast (approx. 6-10AM).
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin at currently prescribed dose

SUMMARY:
Wide variability in the antiplatelet effects of aspirin may lead to recurrent thromboembolic events. Several pilot studies have suggested potential benefits of taking aspirin at bedtime rather than in the morning. The primary objective of this study is to examine whether aspirin administration at bedtime versus in the morning provides a superior reduction in the incidence of major adverse cardiovascular events among patients with or without established atherosclerotic cardiovascular disease, who are already taking aspirin.

DETAILED DESCRIPTION:
The study is a pragmatic, registry-based, open-label, randomized controlled trial combining the utilization of the Danish nationwide health registries and the official Danish electronic letter system (Digital Post/eBoks) into an innovative, decentralized trial requiring no study visits from participants. The nationwide health registries will be used for identification of potential participants and data collection, including baseline information and follow-up data, while the electronic letter system will be used for sending recruitment letters and communicating with participants. Study participants will provide electronic informed consent from home before inclusion and randomization.

The trial will include patients currently in aspirin treatment regardless of the presence or absence of established cardiovascular disease. Participants will be randomized 1:1 to either aspirin administration at bedtime or in the morning. The trial is event-driven.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Current chronic treatment with aspirin (as recorded in the Danish National Prescription Registry and confirmed by the participant via questionnaire)
* Signed informed consent

Exclusion Criteria:

* There are no exclusion criteria for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32706 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Composite of hospitalization for myocardial infarction, hospitalization for stroke, coronary revascularization, or cardiovascular death | Up to 3 years

SECONDARY OUTCOMES:
Hospitalization for myocardial infarction | Up to 3 years
Hospitalization for stroke | Up to 3 years
Coronary revascularization | Up to 3 years
Cardiovascular death | Up to 3 years
All-cause death | Up to 3 years

OTHER OUTCOMES:
Bleeding episode requiring hospitalization | Up to 3 years
Hospitalization for intracranial hemorrhage | Up to 3 years
Hospitalization for gastrointestinal hemorrhage | Up to 3 years
Hospitalization for unstable angina | Up to 3 years
Any arterial revascularization | Up to 3 years
Any venous thromboembolism | Up to 3 years
Time of day of hospitalization for myocardial infarction | Up to 3 years
Time of day of hospitalization for stroke | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Manan Pareek, MD, PhD, Principal Investigator — Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Department of Cardiology, Copenhagen University Hospital - Herlev and Gentofte, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Baseline and endpoint data will be collected from Danish administrative health registries, which are subject to Danish legislation and can only be made available to a third party under certain conditions. Please contact the sponsor in case of any inquiries.